CLINICAL TRIAL: NCT00006447
Title: Supporting Traumatic Brain Injury (TBI) Caregivers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-0106; 5R01HD036075-02 (NIH)
Record Dates: First submitted 2000-11-04; First posted 2000-11-06 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2011-05

CONDITIONS: Traumatic Brain Injuries
Keywords: Brain Injuries; Trauma; Caregivers; Burden and Dependency; Rehabilitation; Support, social; Information System; Information Resources (PT); Disability, persons with
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Wounds and Injuries

INTERVENTIONS:
Procedure: Social Support

SUMMARY:
This randomized trial tested a 6 month intervention of computer network vs a control group (standard care) to improve quality of life and health status for traumatic brain injury (TBI) patients and their caregivers. The network, termed the Trauma Recovery Support System (TRSS), consisted of a central computer system connected via modem to a personal computer in the caregiver's home. Users could access via the Internet special modules and communication services to help them cope with their new roles as caregivers and with accompanying social isolation. These modules were an on-line discussion group, an "ask an expert questions" function, a database of previously asked questions with answers, a database of community resources, and a reference library.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) has long-term and often devastating impacts on a family. The spouse or partner caring for an individual with TBI experiences significant emotional distress, and psychological and physical morbidity. Clinical experience indicates that patients with strong family support progress further than those without family involvement. There is strong evidence that support provided to caregivers improves their well being, as well as that of the care recipient. The trial was designed to lessen her morbidity, improve her support for the TBI partner, and improve recovery of the TBI person.

The effectiveness of a newly developed Trauma Recovery Support System (TRSS) was evaluated using a randomized controlled experimental design. Sixty-four patient/caregiver pairs were recruited, and those (randomly) assigned to the experimental group received access to the centralized TRSS via a personal computer in their homes including access via Internet to special modules and communication services to help them cope with their new roles as caregivers and with accompanying social isolation. Modules consist of an on-line discussion group, an "ask an expert questions" function, a database of previously asked questions with answers, a database of community resources, and a reference library. Controls received standard care. All participants (experimental and control) were interviewed at 0, 3, and 6 months from time of patient discharge, initially in person and later by phone to evaluate the status of the caregiver (quality of life and health status) and TBI patient recovery. Sociodemographic and other background data was collected.

ELIGIBILITY:
Inclusion Criteria:

* Male/female pairs (both at least 18 years of age), where male is recovering from traumatic brain injury (Ranchos Los Amigos Scale class of 1-8) and female spouse/partner is the caregiver

Exclusion Criteria:

* Caregiver (female) not able to read and write English well enough to answer review's questions
* Patients cared for by children, siblings or parents (as opposed to spouse/partner)
* Patients discharged to locations other than home
* Female patients with male caregivers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 1997-09; Primary Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armando James Rotondi — University of Pittsburgh, Dept of Anesthesiology & CCM